CLINICAL TRIAL: NCT07380568
Title: The Effect of Preoperative Oral Melatonin on Postoperative Pain Control After Cesarean Section: A Dose Comparison Study
Brief Title: Melatonin on Post Operative Pain After CS
Acronym: CS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Taghreed Elshahat Sakr, lecturer of anesthesia, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: RC.3.9.2025
Record Dates: First submitted 2025-12-28; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pain Management; Pain After Surgery; Cesarean Section Pain
Keywords: melatonin and pain after C.S
MeSH Terms: conditions — Agnosia | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I: (5 mg melatonin) (Active Comparator)
  Interventions: Drug: Melatonin 5 mg
- Group II: (10 mg melatonin) (Active Comparator)
  Interventions: Drug: Melatonin 10 mg
- Group III: (Placebo) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin 5 mg — Group I: (5 mg melatonin): Participants will receive 5 mg of oral melatonin 1 hours before the cesarean section.
  Arms: Group I: (5 mg melatonin)
Drug: Melatonin 10 mg — Group II: (10 mg melatonin): Participants will receive 10 mg of oral melatonin 1 hours before the cesarean section.
  Arms: Group II: (10 mg melatonin)
Drug: Placebo — Group III: (Placebo): Participants will receive an identical placebo tablet 1 hours before the cesarean section.
  Arms: Group III: (Placebo)

SUMMARY:
The goal of this clinical trial is to learn if melatonin will decrease pain after C.S. The main questions it aims to answer are:

Does melatonin lower the number of times participants need to use a rescue analgesia? What medical problems do participants have when taking melatonin? Researchers will compare different doses of melatonin to see the ideal dose to decrease pain after C.S.

Participants will:

Take melatonin 30 min before C.S and will be observed for 24 hours for pain and consumption of other analgesia

ELIGIBILITY:
Inclusion Criteria:

* - Women aged 18-40 years.
* Scheduled for elective cesarean section.
* Ability to provide informed consent.

Exclusion Criteria:

* Known hypersensitivity to melatonin or opioids
* Chronic use of analgesics, sedatives, or antidepressants.
* History of sleep disorders or psychiatric illness.
* Complicated pregnancies (e.g., preeclampsia, gestational diabetes).
* Body mass index (BMI) > 35 kg/m².
* Emergency cesarean sections.
* Severe systemic diseases (e.g., liver or kidney dysfunction).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity measured using the VAS (Visual Analogue Scale) | 2, 6, 12, and 24 hours post-surgery.
  it typically consists of a 100 mm straight line with descriptive anchors at each end representing the extremes of the sensation (for example, "no pain" at one end and "the most severe pain imaginable" at the other). Respondents indicate their experience by marking a point on the line, and the distance from the lower anchor is measured and recorded as a continuous variable

SECONDARY OUTCOMES:
first rescue analgesia | the first 24 hours post operative
  Time to first request for analgesia postoperatively
Total opioid consumption | the first 24 hours post operative
  amount of opioid requested by the patient
Incidence of adverse effects | first 24 hours post operative
  such as nausea, vomiting, headache, dizziness, sedation
Time to first ambulation post-surgery | first 24 hours post operative
  first movement by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University Hospital, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No